CLINICAL TRIAL: NCT06096714
Title: Addictive Threshold of Nicotine
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000036324; 2U54DA036151-11 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Smoking Addiction
MeSH Terms: interventions — Nicotine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine (Active Comparator): Adaptation Session followed by 4 Test Days. The Adaptation Session will familiarize the participants with study procedures. In each Test Day, a different nicotine dose (0.1, 0.05, 0.025, and 0.0125 mg nicotine/pulse) will be compared to saline for nicotine discrimination, subjective effects, and reinforcement. Participants will first sample the assigned nicotine dose and saline, followed by 4 trials to test their ability to discriminate it from saline. This will be followed by 4 Choice trials where participants will be able to choose between nicotine (at the session-assigned dose) or saline (A or B).
  Interventions: Drug: Nicotine; Other: Saline
- saline (Placebo Comparator): Subjects will have sample A and B, one being nicotine and one being saline. The doses will be blinded from PI, subject and staff. The subject must choose A or B for the next ten choices.
  Interventions: Drug: Nicotine; Other: Saline

INTERVENTIONS:
Drug: Nicotine — Nicotine will be infused using a pump.
Other: Saline — Saline with be used to compare Nicotine, Saline will be infused using a pump

SUMMARY:
To determine the nicotine threshold dose(s) for discrimination, subjective-rewarding effects, -and reinforcement in smokers with different levels of dependence.

DETAILED DESCRIPTION:
The purpose of this project is to determine the nicotine threshold dose(s) for discrimination, subjective-rewarding effects, and reinforcement in smokers with different levels of dependence. Participants will have an Adaptation Session followed by 4 Test Days. The Adaptation Session will familiarize the participants with study procedures. In each Test Day, a different nicotine dose (0.1, 0.05, 0.025, and 0.0125 mg nicotine/pulse) will be compared to saline for nicotine discrimination, subjective effects, and reinforcement. Participants will first sample the assigned nicotine dose and saline, followed by 4 trials to test their ability to discriminate it from saline. This will be followed by 4 Choice trials where participants will be able to choose between nicotine (at the session-assigned dose) or saline to be administered by the research staff.

Reinforcement will be assessed with the percentage of nicotine choices during the Choice trials. The discrimination is the percentage of correctly identified nicotine and saline infusions. Rewarding effects will be assessed with the "Pleasurable Effects" composite score of the Drug Effects Questionnaire (DEQ).

ELIGIBILITY:
Inclusion Criteria:

* to contact their primary care provider when necessary.
* Adults, aged 21 to 59 years. Individuals less than 21 will be excluded because the minimum age for purchasing tobacco products is 21 in our state. The upper age is set at 59 because there are no previous IV nicotine studies that enrolled smokers over the age of 59.
* Smoking at least for one year and more frequently than once a week, smoking status confirmed with a semi-quantitative urine nicotine test. Smokers will be stratified based on the level of dependence, assessed with the FTND scores (Heatherton et al. 1991) (low or no dependence 4 and moderate or high level of dependence 5.
* In good health as verified by medical history, screening examination, and screening laboratory tests.
* For women, report using acceptable birth control methods.

Exclusion Criteria:

* History of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the participant to be in the study
* regular current use of certain psychotropic medications (such as mood stabilizers, antipsychotics, or anxiolytics being prescribed to treat bipolar disorder, psychosis or anxiety spectrum disorders, respectively)
* current untreated alcohol or substance use disorder for any other recreational or prescription drugs other than nicotine
* for women, pregnant as determined by pregnancy screening, or breastfeeding
* seeking (or undergoing) treatment for tobacco dependence or smoking.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
correctly identifying nicotine | up to 8 weeks
  Reinforcement will be assessed with the percentage of nicotine doses chosen during the Choice trials (out of 16), 4 choices per day over four days.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No